CLINICAL TRIAL: NCT02513953
Title: Endometrioma in Layers of Brot ad Ligament in Left Adnexa
Brief Title: Case Report of Endometrioma in Layers of Broad Ligament.
Acronym: mesosalpinx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruby Hall IVF and Endoscopy Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endometriosis
Record Dates: First submitted 2015-07-28; First posted 2015-08-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Theca Lutein Cyst of Left Ovary
Keywords: Endometriosis; Mesosalpinx; Broad Ligament; Laparoscopy
MeSH Terms: conditions — Endometriosis | interventions — Laparoscopy; Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endometriosis (Experimental): Four port laparoscopy by way of intervention was needed for convenience in aspirating the cystic fluid and reversal of the cyst wall taking care not to destroy the normal ovarian tissue to minimize loss of ovarian reserve
  Interventions: Procedure: Laparoscopic

INTERVENTIONS:
Procedure: Laparoscopic — Four Port Laparoscopic cystectomy
  Other Names: cystectomy

SUMMARY:
Objective:To present an extremely rare site of occurrence of endometriotic cyst in the layers of Broad Ligament.

Patient:A 32 yrs.old woman,married 4 yrs.,presented to OB-GY Dept.with acute,gnawing pain in lower abdomen and history of sub-fertility.Diagnostic Laparoscopy and pelvic ultrasound were performed in emergency.Oblong cyst structure,41x21x23mm in the left adnexa,away from ovary and uterus was identified and excised by Four Port laparoscopic interventional surgery.

DETAILED DESCRIPTION:
Endometriosis is the second most common finding in the pelvis of females in their reproductive age, frequently associated with primary infertility. Endometrioma, within layers of broad ligament has been reported, but only in four cases, so far.

Contributing factors in the etiopathogenesis of endometriosis and endometriomas are retrograde menstrual flow, metaplasia, genetic predisposition, lymphatic/ vascular distribution, immune dysfunction and environmental influences. Etiopathogenesis of endometriosis is still poorly understood, the main theories being embryonic, migratory and immunologic. Embryonic theories suggest that endometriosis develops from the remnants of wolffian ducts or the Mullerian ducts or may develop from the metaplasia of the peritoneal or the ovarian tissue. Migratory theories suggest transportation of endometrial tissue to distant places via fallopian tubes or, lymphovascular structure and subsequent implantation as the cause of endometriosis. Immunologic theory implies that altered immune response may help in ectopic endometrial implantation. However, all these mechanisms may act synergistically and not in exclusion of each other. Endometrial alterations in the eutopic endometrium have also been demonstrated in women with endometriosis. These alterations involve progesterone receptors co - activator, Hic - 5 resulting in resistance to progesterone. Endometriosis commonly involves ovaries, POD, uterosacral ligaments and rectovaginal septum, all within the pelvis. This accounts for the retrograde menstruation being the most popular theory of pathogenesis for endometriosis. But endometriosis may develop at many unusual locations incl. abdominal wall, urinary system, gastrointestinal system, thorax, inguinal canal, large muscular or in few cases, within the layers of broad ligament.

Endometriosis, within the layers of broad ligament presents with classical symptoms of pelvic endometriosis, triad of chronic pelvic pain, dysmenorrhea and dyspareunia. Our patient, under reporting, presented with throbbing pain in lower abdomen. Other descriptions of pain being gnawing pain or dragging pain to the legs. Compared to women with superficial endometriosis, those with deep disease are more likely to report dyschezia. All the four cases of endometriosis of broad ligament reported so far, had one or more of these symptoms, the most common being episodic or continuous in low abdomen. All these cases reported were 27 - 34yrs old. Although, endometriosis is strongly associated with infertility no association between broad ligament endometrioma and infertility has been reported so far. Previously reported cases have been either parous or nulliparous females not desirous of childbearing, our patient under reporting, is the first case being reported as a female presenting with subfertility. This association needs to be explored in future because apart from localized endometrioma, there were no other locations of endometriosis anywhere in the pelvis, in ovarian fossa, in POD or anywhere else. Could it be that implantation is the prerequisite in endometriomas causing infertility? Complete excision of cyst wall is preferred over drainage and ablation. The female patient was posted for operative laparoscopy in the post - menstrual period. Four port laparoscopy was preferred to visualize oblong cystic structure, measuring 4x3cms within the layers of left mesosalpinx. A small incision was applied on the most prominent part of the cyst on the posterior leaf of mesosalpinx and thick chocolate fluid was suctioned out. Cystectomy was performed, dissecting the cyst wall from the leaves of mesosalpinx, using harmonic. Posterior leaf of mesosalpinx was repaired with three interrupted sutures using vicryl no.1. Through peritoneal lavage with normal saline was given. Patient was discharged on the same day after uncomplicated post - operative period.

ELIGIBILITY:
Inclusion Criteria:Sub-fertile women with confirmed diagnosis of pelvic endometriosis.

-

Exclusion Criteria:women with Pelvic inflammatory disorders and other forms of benign cysts.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
cystectomy of endometrioma in layers of Broad Ligament | Forty five minutes.
  Laparoscopic surgery under general anaesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Parinazz Parhar, MBBS, Study Chair — Ruby Hall Clinic